CLINICAL TRIAL: NCT03091504
Title: Evaluation on the Efficacy of Bronchodilator Nebulization Via High Flow Nasal Cannula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: People's Hospital of Xinjiang Uygur Autonomous Region (Other)
Responsible Party: Principal Investigator, Jie Li, Principal Investigator, Rush University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BDTHFNC01
Record Dates: First submitted 2017-03-15; First posted 2017-03-27 (Actual); Last update posted 2018-04-04 (Actual); Status verified 2018-04

CONDITIONS: High Flow Nasal Cannula
MeSH Terms: interventions — Albuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Albuterol via High flow nasal cannula (Experimental): Enrolled patients inhale bronchodilator (Albuterol Sulfate) with different concentration via High flow nasal cannula, prepared albuterol concentrations are 0.5mg, 1.0mg, 2.0mg and 4.0mg, patients will be assessed by spirometry after each concentration until bronchodilator response is positive and does not improve after the next dose.
  Interventions: Device: High flow nasal cannula; Drug: Albuterol Sulfate

INTERVENTIONS:
Device: High flow nasal cannula — High flow nasal cannula is a soft and flexible nasal prongs with adjustable head strap fits over the patient's ears, it delivers a broad variety of gas flows directly into the nares without gas jetting.
  Other Names: Optiflow, Fisher Paykel
Drug: Albuterol Sulfate — Albuterol is a short acting inhaled bronchodilator
  Other Names: Ventolin

SUMMARY:
High-humidity nasal cannula (HFNC) has been shown to be effective in improving oxygenation and avoiding intubation in multiple randomized control trials, it is also suitable and feasible for long term use. Aerosol delivery via HFNC will minimize interruptions and improve patient compliance, bench study and radionuclide imaging study done in healthy volunteers demonstrated that aerosol can be effectively delivered using HFNC. This study aims to evaluate the efficacy of bronchodilator delivered via HFNC in chronic pulmonary obstructive disease or asthma patients.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease or asthma patients who have positive response in bronchodilator test will be consented and enrolled, patients come back for the second bronchodilator assessment within one to three days after the initial bronchodilator test. Albuterol with different concentration will be provided to the patients via HFNC, patients will be assessed by spirometry after each concentration until bronchodilator response is positive and does not improve after the next dose.

ELIGIBILITY:
Inclusion Criteria:

* Diagnose with COPD or asthma
* Bronchodilator test is positive (According to ATS guidelines, FEV1 change from initial more than 12% and FEV1 absolute change more than 200 mL);
* Age > 18yrs and < 90yrs

Exclusion Criteria:

* Recent pulmonary exacerbation
* Mental disease
* Uncooperative
* Reluctant to participate
* Patients who are unable to come back to get the second spirometry within three days
* Contraindicated to Albuterol (Ventolin, GSK)

  * Rest HR > 100 beats/min
  * Serum K+ < 2.8 mmol/L

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-09-04 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
FEV1 change from initial | 30-60 mins
  FEV1 abs Δ: post FEV 1 - pre FEV1 and FEV1 %Δinit: (post FEV1 - pre FEV1)/pre FEV1 × 100

SECONDARY OUTCOMES:
Breath sound | 30-60 mins
  Wheezing
Heart rate | 30-60 mins
  The number of heart beats per minute
Respiratory rate | 30-60 mins
  About 4,630,000 results (0.68 seconds)
  Search Results
  The number of breaths per minute
Side effects | 30-60 mins
  Tremor

CONTACTS AND LOCATIONS:
Overall Officials: Minghua Zhao, MD, Principal Investigator — People's Hospital of Xinjiang Uygur Autonomous Region
Locations (1):
- People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dailey PA, Harwood R, Walsh K, Fink JB, Thayer T, Gagnon G, Ari A. Aerosol Delivery Through Adult High Flow Nasal Cannula With Heliox and Oxygen. Respir Care. 2017 Sep;62(9):1186-1192. doi: 10.4187/respcare.05127. Epub 2017 Jun 6. PMID 28588117
- [Background] Reminiac F, Vecellio L, Heuze-Vourc'h N, Petitcollin A, Respaud R, Cabrera M, Pennec DL, Diot P, Ehrmann S. Aerosol Therapy in Adults Receiving High Flow Nasal Cannula Oxygen Therapy. J Aerosol Med Pulm Drug Deliv. 2016 Apr;29(2):134-41. doi: 10.1089/jamp.2015.1219. Epub 2015 Jul 21. PMID 26196740
- [Background] Dugernier J, Hesse M, Jumetz T, Bialais E, Roeseler J, Depoortere V, Michotte JB, Wittebole X, Ehrmann S, Laterre PF, Jamar F, Reychler G. Aerosol Delivery with Two Nebulizers Through High-Flow Nasal Cannula: A Randomized Cross-Over Single-Photon Emission Computed Tomography-Computed Tomography Study. J Aerosol Med Pulm Drug Deliv. 2017 Oct;30(5):349-358. doi: 10.1089/jamp.2017.1366. Epub 2017 May 2. PMID 28463044
- [Background] Reminiac F, Vecellio L, Loughlin RM, Le Pennec D, Cabrera M, Vourc'h NH, Fink JB, Ehrmann S. Nasal high flow nebulization in infants and toddlers: An in vitro and in vivo scintigraphic study. Pediatr Pulmonol. 2017 Mar;52(3):337-344. doi: 10.1002/ppul.23509. Epub 2016 Jul 8. PMID 27392199
- [Background] Morgan SE, Mosakowski S, Solano P, Hall JB, Tung A. High-Flow Nasal Cannula and Aerosolized beta Agonists for Rescue Therapy in Children With Bronchiolitis: A Case Series. Respir Care. 2015 Sep;60(9):e161-5. doi: 10.4187/respcare.03996. Epub 2015 Jun 23. PMID 26106204
- [Background] Baudin F, Buisson A, Vanel B, Massenavette B, Pouyau R, Javouhey E. Nasal high flow in management of children with status asthmaticus: a retrospective observational study. Ann Intensive Care. 2017 Dec;7(1):55. doi: 10.1186/s13613-017-0278-1. Epub 2017 May 22. PMID 28534235